CLINICAL TRIAL: NCT03956615
Title: sdAb-based Targeted Radionuclide Therapy of Multiple Myeloma: a Feasibility Study
Brief Title: sdAb-based TRNT of Multiple Myeloma: a Feasibility Study
Acronym: MUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Stichting tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UZBRU_MUM
Record Dates: First submitted 2019-04-18; First posted 2019-05-21 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinically Suspected or Pathologically Confirmed Multiple Myeloma. (Other): Patients with a clinically suspected or pathologically confirmed multiple myeloma.
  Interventions: Other: Blood sampling and bone marrow analysis

INTERVENTIONS:
Other: Blood sampling and bone marrow analysis — Bone marrow sample analysis. A blood sampling of maximally 10 ml by venous puncture (serum)

SUMMARY:
This study aims to show that antiidiotypic sdAb are a new, sensitive, specific and non-invasive tool for imaging and therapeutic purposes and provides a rationale for their clinical evaluation as a personalized treatment option for MM patients expressing surface paraprotein.

ELIGIBILITY:
Inclusion Criteria:

Patients will only be included in the study if they meet all of the following criteria:

* Patients who have given informed consent
* Patients at least 18 years old
* Patients scheduled to undergo bone marrow sampling in clinical routine because of a clinically suspected or pathologically confirmed multiple myeloma.

Exclusion Criteria:

Patients will not be included in the study if one of the following criteria applies:

* Patients who cannot communicate reliably with the investigator
* Patients who are unlikely to cooperate with the requirements of the study
* Patients at increased risk of death from a pre-existing concurrent illness
* Patients who participated already in part I of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Keyaerts, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinically Suspected or Pathologically Confirmed Multiple Myeloma.: Only 1 arm/group in this trial - Patients with a clinically suspected or pathologically confirmed multiple myeloma.
Period: Overall Study
Arm/Group | Clinically Suspected or Pathologically Confirmed Multiple Myeloma.
Started | 10
Completed | 3
Not Completed | 7
Not completed — No multiple myeloma confirmed | 2
Not completed — Assessment of membrane-expressed ideotypic paraprotein not possible due to low CD38 signals | 1
Not completed — No expression of ideotypic paraprotein on membrane | 2
Not completed — Not selected for sdAb generation, due to limitation of total number to 3 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Clinically Suspected or Pathologically Confirmed Multiple Myeloma.
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 10

OUTCOME MEASURES:

1. Primary Outcome: Fraction of Patients (n=3) for Whom a sdAb Could be Generated That Binds to the Idiotype of the Paraprotein.
Description: Reporting of the relative amount of patients for whom such sdAb could be successfully obtained
Time Frame: Within 2 years after study completion
Population: Out of 10 patients included, three patients with confirmed surface Ig expression were selected for sdAb generation.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With a Clinically Suspected or Pathologically Confirmed Multiple Myeloma.: Only 1 arm/group in this trial
Arm/Group | Patients With a Clinically Suspected or Pathologically Confirmed Multiple Myeloma.
Number analyzed (Participants) | 3
Participants | 2

2. Primary Outcome: Amount of Paraprotein-targeting sdAbs Generated Per Patient
Description: Absolute amount of unique sdAbs obtained per patient
Time Frame: Within 2 years after study completion
Population: Per participant, the number of different SdAb generated are reported.
Measure: Number; unit: unique sdAbs
Arm/Group | Patients With a Clinically Suspected or Pathologically Confirmed Multiple Myeloma.
Number analyzed (Participants) | 3
unique sdAbs
  number of different SdAb for subject 1: number analyzed (Participants) | 1
  number of different SdAb for subject 1 | 14
  number of different SdAb for subject 2: number analyzed (Participants) | 1
  number of different SdAb for subject 2 | 0
  number of different SdAb for subject 5: number analyzed (Participants) | 1
  number of different SdAb for subject 5 | 20

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Patients With a Clinically Suspected or Pathologically Confirmed Multiple Myeloma.
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT03956615/Prot_SAP_000.pdf